CLINICAL TRIAL: NCT07353463
Title: Shanghai Clinical Cohort - Parkinson's Disease (Reserve)
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Huashan Hospital (Other); Shanghai Yangzhi Rehabilitation Hospital (Unknown); Longhua Hospital (Other); Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: Parkinson's Disease Cohort; SHDC2025CCS043 (Other Grant/Funding Number: Shanghai Shenkang Hospital Development Center)
Record Dates: First submitted 2025-11-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease (PD); Multiple System Atrophy
Keywords: observational cohort study; multimodal data; subtyping; long-term monitoring
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The study will retain multiple types of biospecimens, including:
  Blood samples (whole blood, serum, plasma, DNA extraction) Saliva samples Cerebrospinal fluid (CSF) (optional, with patient consent)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease Cohort: This cohort will include approximately 600 patients diagnosed with Parkinson's disease according to established Chinese diagnostic criteria. Participants will undergo standardized clinical assessments of motor and non-motor symptoms, neuroimaging (MRI, optional PET/SPECT), electrophysiological recordings, and collection of biospecimens (blood, saliva, optional CSF). Longitudinal follow-up will be conducted every 6 months to monitor disease progression and treatment response.
- Multiple System Atrophy Cohort: This cohort will include approximately 100 patients with clinically diagnosed or probable multiple system atrophy, based on Chinese expert consensus criteria. Participants will undergo comprehensive clinical evaluation, neuroimaging, electrophysiological testing, and biospecimen collection (blood, saliva, optional CSF). Regular follow-up every 6 months will capture disease progression, functional decline, and potential biomarkers.

SUMMARY:
The goal of this observational cohort studyis to establish a high-quality clinical cohort of Parkinson's disease (PD) and multiple system atrophy (MSA) patients in Shanghai, in order to improve early diagnosis, precise subtyping, disease monitoring, and to provide a resource for translational research and novel therapy development.

The main questions it aims to answer are:

* Can multimodal data (clinical, imaging, electrophysiology, biospecimens, and genetics) help identify early biomarkers for PD and MSA?
* Can precise subtyping and long-term monitoring predict disease progression and therapeutic response? Researchers will compare 600 PD patients and 100 MSA patients to evaluate differences in clinical features, biomarkers, imaging, and prognosis.

Participants will:

* Provide informed consent and complete baseline demographic and medical history collection.
* Undergo standardized clinical evaluations, including motor and non-motor symptom scales, cognitive and quality-of-life assessments.
* Provide biological samples (blood, saliva, optional CSF).
* Receive brain imaging (MRI, optional PET/SPECT) and electrophysiological recordings (EEG, fNIRS).
* Participate in longitudinal follow-up visits every 6 months for repeat assessments.

This study will create a sustainable, multicenter, and sharable cohort platform to support early identification, personalized intervention, and therapeutic development for neurodegenerative diseases

ELIGIBILITY:
* Inclusion Criteria for Clinical PD Group:

  1. Patients with a clinical diagnosis of Parkinson's disease (PD) according to the _Chinese Diagnostic Criteria for Parkinson's Disease (2016 edition)_.
  2. Willingness to undergo biospecimen collection, including cerebrospinal fluid (optional), blood, and saliva, and to complete neuroimaging examinations (MRI, PET/SPECT) and disease-specific clinical assessments.
  3. Provision of written informed consent
* Inclusion Criteria for Clinical MSA Group:

  1. Patients with a clinical diagnosis or clinically probable multiple system atrophy (MSA) according to the Chinese Expert Consensus on the Diagnostic Criteria for MSA (2022).
  2. Willingness to undergo biospecimen collection, including cerebrospinal fluid (optional), blood, and saliva, and to complete neuroimaging examinations (MRI, PET/SPECT) and disease-specific clinical assessments.
  3. Provision of written informed consent.
* Exclusion Criteria for All Participants:

  1. Patients with an unclear or uncertain diagnosis.
  2. History of stroke, head trauma, hydrocephalus, brain tumor, intracranial hypertension, or intracranial surgery.
  3. Evidence of intracranial organic lesions on CT/MRI.
  4. Severe anxiety, depression, or schizophrenia.
  5. Severe comorbidities involving the heart, lungs, liver, kidneys, endocrine system, or hematological system.
  6. Presence of aphasia, severe dysarthria, or other conditions that significantly impair clinical assessments.
  7. Anticipated poor compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with Parkinson's disease (PD) and multiple system atrophy (MSA) recruited from outpatient and inpatient clinics at Ruijin Hospital and collaborating tertiary medical centers in Shanghai. Approximately 600 clinically diagnosed PD patients and 100 clinically diagnosed or probable MSA patients will be enrolled. All participants must meet established Chinese diagnostic criteria, agree to provide biospecimens (blood, saliva, optional CSF), undergo neuroimaging and electrophysiological testing, and complete standardized clinical assessments. Patients with unclear diagnoses, significant comorbidities, or poor compliance will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in motor symptom severity assessed by MDS-UPDRS Part III | From baseline through 6-month and 12-month follow-up assessments
  Motor symptom severity will be assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS Part III; range 0-132, higher scores indicate worse motor impairment). The primary outcome is the change from baseline score.
Change from baseline in Hoehn & Yahr stage | From baseline through 6-month and 12-month follow-up assessments
  Disease severity will be assessed using the Hoehn & Yahr staging scale, which classifies Parkinson's disease severity on a scale from Stage 1 to Stage 5, with higher stages indicating more advanced disease. The secondary outcome is the change in Hoehn & Yahr stage from baseline.
Change from baseline in Brief Pain Inventory (BPI) pain severity score | From baseline through 6-month and 12-month follow-up assessments
  Pain severity will be assessed using the Brief Pain Inventory (BPI) pain severity subscale, with scores ranging from 0 to 10. Higher scores indicate more severe pain. The secondary outcome is the change from baseline in BPI pain severity score.
Change from baseline in REM Sleep Behavior Disorder Questionnaire-Hong Kong (RBDQ-HK) score | From baseline through 6-month and 12-month follow-up assessments
  REM sleep behavior disorder symptoms will be assessed using the REM Sleep Behavior Disorder Questionnaire-Hong Kong (RBDQ-HK), with total scores ranging from 0 to 100. Higher scores indicate more severe RBD symptoms. The secondary outcome is the change from baseline in RBDQ-HK score.
Change from baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLSS) score | From baseline through 6-month and 12-month follow-up assessments
  Restless legs syndrome symptom severity will be assessed using the International Restless Legs Syndrome Study Group Rating Scale (IRLSS), with scores ranging from 0 to 40. Higher scores indicate more severe symptoms. The secondary outcome is the change from baseline in IRLSS score.
Change from baseline in University of Pennsylvania Smell Identification Test (UPSIT) score | From baseline through 6-month and 12-month follow-up assessments
  Olfactory function will be assessed using the University of Pennsylvania Smell Identification Test (UPSIT), with scores ranging from 0 to 40. Lower scores indicate worse olfactory function. The secondary outcome is the change from baseline in UPSIT score.
Change from baseline in Scales for Outcomes in Parkinson's Disease-Autonomic (SCOPA-AUT) score | From baseline through 6-month and 12-month follow-up assessments
  Autonomic dysfunction will be assessed using the Scales for Outcomes in Parkinson's Disease-Autonomic (SCOPA-AUT), with total scores ranging from 0 to 69. Higher scores indicate more severe autonomic dysfunction. The secondary outcome is the change from baseline in SCOPA-AUT score.
Change from baseline in Epworth Sleepiness Scale (ESS) score | From baseline through 6-month and 12-month follow-up assessments
  Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (ESS), with scores ranging from 0 to 24. Higher scores indicate greater daytime sleepiness. The secondary outcome is the change from baseline in ESS score.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) score | From baseline through 6-month and 12-month follow-up assessments
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), with total scores ranging from 0 to 21. Higher scores indicate poorer sleep quality. The secondary outcome is the change from baseline in PSQI score.
Change from baseline in Hamilton Anxiety Rating Scale (HAMA) score | From baseline through 6-month and 12-month follow-up assessments
  Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HAMA), with total scores ranging from 0 to 56. Higher scores indicate more severe anxiety. The secondary outcome is the change from baseline in HAMA score.
Change from baseline in Hamilton Depression Rating Scale-17 (HAMD-17) score | From baseline through 6-month and 12-month follow-up assessments
  Depressive symptoms will be assessed using the 17-item Hamilton Depression Rating Scale (HAMD-17), with total scores ranging from 0 to 52. Higher scores indicate more severe depressive symptoms. The secondary outcome is the change from baseline in HAMD-17 score.
Change from baseline in Non-Motor Symptoms Scale (NMSS) total score | From baseline through 6-month and 12-month follow-up assessments
  Non-motor symptom burden will be assessed using the Non-Motor Symptoms Scale (NMSS), with total scores ranging from 0 to 360. Higher scores indicate greater severity of non-motor symptoms. The secondary outcome is the change from baseline in NMSS total score
Change from baseline in Montreal Cognitive Assessment (MoCA) score | From baseline through 6-month and 12-month follow-up assessments
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), with scores ranging from 0 to 30. Lower scores indicate worse cognitive performance. The secondary outcome is the change from baseline in MoCA score.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No